CLINICAL TRIAL: NCT01837186
Title: Incidence, Risk Factors and Outcome of Empyema Following Pneumonectomy for Non Small Cell Lung Cancer (NSCLC)
Brief Title: Empyema Following Pneumonectomy for Non Small Cell Lung Cancer (NSCLC)
Status: Completed | Type: Observational
Sponsor: University Hospital, Gasthuisberg (Other)
Responsible Party: Principal Investigator, Johnny Moons, Datamanager Thoracic Surgery, University Hospital, Gasthuisberg
Other Study IDs: EMPY2013
Record Dates: First submitted 2013-04-15; First posted 2013-04-23 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Non Small Cell Lung Cancer; Lung Cancer
Keywords: Surgery; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- EFP: Empyema following pneumonectomy
- nEFP: No empyema following pneumonectomy

SUMMARY:
Empyema following pneumonectomy for Non Small Cell Lung Cancer (NSCLC) is a known problem that occurs in about 2% of pneumonectomy patients.

DETAILED DESCRIPTION:
The development of an empyema following pneumonectomy is a devastating complication, especially if associated with an underlying fistula. Whilst the perioperative mortality of pneumonectomy overall is now less than 5%, this rises to around 25% when complicated by empyema, and about 50% when associated with fistula. In addition, there is the morbidity and social cost of long-term drainage, chronic sepsis and often multiple operations.

ELIGIBILITY:
Inclusion Criteria:

* Pneumonectomy for NSCLC

Exclusion Criteria:

* Pneumonectomy for other reasons (infectious pathology, trauma, mesothelioma, ...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive pneumonectomies for Non Small Cell Lung Cancer (NSCLC) from the University Hospital Leuven from 1996 till 2012
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2012-01; Primary Completion 2012-09 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Overall survival | 5 years from surgery
  overall 5-year survival after empyema following pneumonectomy

SECONDARY OUTCOMES:
incidence rate | 1 and 5 years from surgery
  incidence of empyema, accompanied with broncho-pleural fistula or not, divided in short term (less than 1 yr postoperatively) and long term (up to 5 years postoperatively) incidence.

OTHER OUTCOMES:
fast track treatment outcome | 5 years from surgery
  over the last 7 years, a new approach - known as 'fast track treatment of Empyema following pneumonectomy (EFP)' is used. We will examine if there is a benificial aspect in this approach, regarding survival en hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Paul De Leyn, PhD; MD, Study Director — UZ Leuven, Dept. Thoracic Surgery; Arnaud Colle, Principal Investigator — University Leuven
Locations (1):
- University Hospital Leuven, Dept. Thoracic Surgery, Leuven, Belgium